CLINICAL TRIAL: NCT00547326
Title: The Effect of Osteopatic Cranial Techniques on the Audiometric and Tympanometric Values in Children Suffering From Otitis Media With Effusion.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics Committee approval denied
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2007/397
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatement with osteopatic cranial techniques
  Interventions: Procedure: treated with osteopatic cranial techniques
- 2 (Placebo Comparator): Treatment with placebo
  Interventions: Procedure: Treatment with placebo

INTERVENTIONS:
Procedure: treated with osteopatic cranial techniques — treated with osteopatic cranial techniques
  Arms: 1
Procedure: Treatment with placebo — Treatment with placebo
  Arms: 2

SUMMARY:
Children with otitis media with effusion will be treated with osteopatic cranial techniques or with a placebo treatment. Before and after the treatment audiometric and tympanometric measures will take place. This procedure will be repeated 3 times, once a week and every session will last for 30-45 minutes. The fourth week, only audiometry and tympanomtry will be done.

ELIGIBILITY:
Inclusion Criteria:

* children between 3 and 7 years old
* Bilateral otitis media with effusion
* Tympanogram type B

Exclusion Criteria:

* ventilation tubes
* Damage of the tympanic membrane
* Operation of the tympanic membrane
* Other illness e.g. Down, craniofacial abnormalities,…

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Audiometric and tympanometric results | directly after every session of treatment (3 times, once a week)

SECONDARY OUTCOMES:
Audiometric and tympanometric results | one week after the last treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: I. Dhooge, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be